CLINICAL TRIAL: NCT06191237
Title: Effect of Environmental Temperature on Vascular Ultrasound Vein Scan Measurements
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Mr Zeeshan Ahmed Consultant vascular Surgeon, University Hospital of Limerick
Other Study IDs: DVS009
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We wish to conduct two vascular ultrasound scans conducting vein measurements in two separate scanning rooms to assess if environmental temperature affects the vein diameter recorded.

DETAILED DESCRIPTION:
Vascular surgeons are guided by vascular ultrasound scans when deciding treatment plans for their patients. In critical limb threatening ischaemia with infrainguinal disease, vein bypass has the best limb salvage and long term survival rates in patients who are appropriately selected. In lower limb "vein mapping", the vein is measured to assess suitability for use as a bypass conduit with the favoured bypass conduit being autologous, ipsilateral vein of good quality and length and a size of >3mm is considered a good conduit.

The research team found one study which explored the effect of room temperature on upper limb vein measurements which was conducted in Singapore. This showed an underestimation of vein size at lower temperatures. We wish to add to the literature and irish research by conducting this study at University Hospital Limerick in order to optimise conditions for vascular assessments and therefore facilitate clinical decision making.

We aim to scan and record vein measurements on the lower limbs of vascular inpatients at University Hospital Limerick who are deemed suitable by the P.I.

Patients will have the ultrasound scan completed twice. The first room will have its temperature recorded and the vein measurements taken.

The second room will be set at a higher temperature which we have defined as being 6-10 degrees greater than ambient room temperature. We will achieve this through use of a portable heater.

We will compare the two recordings to assess if there is a difference in the diameter of the vein measured in the warmer room versus the standard room.

The importance of this is to assess the impact of environmental factors on vascular ultrasound scan results, therefore impacting on patient outcomes by use of the most suitable bypass conduit.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at University Hospital Limerick under the care of a Vascular Consultant
* Aged 18 years and above
* Deemed suitable for two vascular ultrasound scans by the P.I

Exclusion Criteria:

* Those unable to give informed consent
* Aged under 18 years
* Patients with varicose veins/venous insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who meet inclusion criteria under the care of a Consultant Vascular Surgeon with no varicose veins/venous insufficiency will have vascular ultrasound vein scans performed and measurements recorded.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Vein diameter measurements in two temperature controlled rooms | 3 months
  Two vascular ultrasound scans will be performed on the lower limb. A defined scanning protocol will be adhered to which will ensure consistency and accuracy.
  During the course of both ultrasound scans, vein measurements will be taken and recorded on the study sheet which will have the participant study identification number, age and gender.
  The second room will be set at a higher temperature which we have defined as being 6-10 degrees greater than ambient room temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Ahmed, FRCS, Principal Investigator — Consultant Vascular Surgeon

IPD SHARING:
Plan to Share IPD: No